CLINICAL TRIAL: NCT01086878
Title: Safety of Cotrimoxazole in HIV- and HAART-exposed Infants in Botswana
Brief Title: Safety of Cotrimoxazole in HIV- and HAART-exposed Infants
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Harvard School of Public Health (HSPH) (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Fogarty International Center of the National Institute of Health (NIH); Harvard Initiative for Global Health (Unknown); The American Society of Tropical Medicine and Hygiene (Other)
Responsible Party: Shahin Lockman, MD, Harvard School of Public Health
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: BHP031; 2P30AI060354-06 (NIH); 3R24TW007988-01S1 (NIH)
Record Dates: First submitted 2010-03-12; First posted 2010-03-15 (Estimated); Last update posted 2011-02-25 (Estimated); Status verified 2011-02

CONDITIONS: Acquired Immunodeficiency Syndrome; Infant, Newborn; Anemia; Neutropenia; HIV Infections
Keywords: Antiretroviral Therapy, Highly Active; Trimethoprim-Sulfamethoxazole Combination; anemia; neutropenia; safety; hematologic toxicity
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Anemia; Neutropenia; HIV Infections | interventions — Trimethoprim, Sulfamethoxazole Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cotrimoxazole (Experimental)
  Interventions: Drug: cotrimoxazole

INTERVENTIONS:
Drug: cotrimoxazole — Daily oral cotrimoxazole suspension from 1 to 6 months of age at the following weight-based doses:
  * less than 5kg: 100mg sulfamethoxazole, 20mg trimethoprim
  * greater than 5kg: 200mg sulfamethoxazole, 40mg trimethoprim
  Other Names: Bactrim; Septrim; Cotrim; Septra; trimethoprim/sulfamethoxazole; trimethoprim-sulfamethoxazole

SUMMARY:
The purpose of this study is to determine if prophylactic cotrimoxazole makes severe anemia or neutropenia more common in infants exposed to maternal HIV and combination antiretroviral therapy.

DETAILED DESCRIPTION:
Each year, more than 2 million children are born to HIV-infected women. The World Health Organization (WHO) recommends that these infants receive cotrimoxazole (CTX) prophylaxis starting at 4-6 weeks of age until the period of infant HIV transmission risk is over, and the infant is known to be HIV-uninfected. There is also increasing interest in studying CTX prophylaxis given to all infants of HIV-infected women at the time of initiation of replacement feeding, regardless of infant HIV infection status, to mitigate the high risk of infant morbidity and mortality associated with formula feeding in the developing world. However, infant in utero exposure to maternal antiretroviral drugs can lead to hematologic toxicities in infants. It is critical to know whether infant CTX prophylaxis exacerbates the hematologic toxicity associated with perinatal ARV exposure. This question, with broad public health implications, has never been studied.

We will study the hematologic toxicity associated with CTX prophylaxis given to infants exposed to maternal HAART in Botswana. We will use existing data from a large cohort that did not receive CTX, and enroll a smaller cohort that does receive CTX according to Botswana national guidelines.

ELIGIBILITY:
Both maternal and infant criteria need to be met:

Maternal Inclusion Criteria:

* documented HIV infection
* taking 3-drug highly active antiretroviral therapy at any point during pregnancy (note: can include 2 NRTI+NNRTI, 2NRTI+PI, or 3 NRTI)
* 21 years of age or older, and able and willing to sign informed consent
* Proof of Botswana Citizenship

Maternal Exclusion Criteria:

* involuntary incarceration

Infant Inclusion Criteria:

* younger than 42 days of age
* able to be brought to regular visits at study clinic until at least 6 months postpartum

Infant Exclusion Criteria:

* known pre-existing birth anomalies resulting in a high probability that the baby will not survive to 6 months
* known hypersensitivity to cotrimoxazole

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 222 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
incidence of severe or life-threatening anemia | between 1 to 6 months of life
  incidence of severe or life-threatening anemia (as defined by DAIDS toxicity tables, 2004) between 1 and 6 month of life

SECONDARY OUTCOMES:
incidence of severe or life-threatening neutropenia | between 1 to 6 months of life
  incidence of severe or life-threatening neutropenia (as defined by DAIDS toxicity tables, 2004) between 1 and 6 month of life
composite severe morbidity and mortality | between 1 and 6 months of life
  Composite of severe morbidity (grade 3 or 4 illnesses, DAIDS toxicity tables, 2004), hospitalization, and mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Shahin Lockman, MD, Principal Investigator — Harvard School of Public Health (HSPH)
Locations (2):
- Botswana (2):
  - Princess Marina Hospital, Gaborone, Gaborone
  - Scottish Livingstone Hospital, Molepolole, Kweneng District

REFERENCES:
- [Derived] Dryden-Peterson S, Jayeoba O, Hughes MD, Jibril H, McIntosh K, Modise TA, Asmelash A, Powis KM, Essex M, Shapiro RL, Lockman S. Cotrimoxazole prophylaxis and risk of severe anemia or severe neutropenia in HAART-exposed, HIV-uninfected infants. PLoS One. 2013 Sep 23;8(9):e74171. doi: 10.1371/journal.pone.0074171. eCollection 2013. PMID 24086319